CLINICAL TRIAL: NCT02954198
Title: Once-daily Regimen With Envarsus® to Optimize Immunosuppression Management and Outcomes in Kidney Transplant Recipients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00059602
Record Dates: First submitted 2016-10-13; First posted 2016-11-03 (Estimated); Results first posted 2019-12-24 (Actual); Last update posted 2019-12-24 (Actual); Status verified 2019-12

CONDITIONS: Immunosuppression
MeSH Terms: interventions — Tacrolimus; Prednisone; Adrenal Cortex Hormones; Methylprednisolone; Mycophenolic Acid; Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tacrolimus + MMF (Active Comparator): Tacrolimus IR BID (5-12ng/mL) + mycophenolate mofetil 1g BID + prednisone x at least 3 months, then converted to Tacrolimus Daily (5 -12ng/mL) + mycophenolate mofetil 1g BID + prednisone x 6 months
  Interventions: Drug: Tacrolimus; Drug: Prednisone; Drug: Mycophenolate mofetil
- Envarsus + Everolimus (Active Comparator): Tacrolimus IR BID (5-12ng/mL) + mycophenolate mofetil 1g BID + prednisone x at least 3 months, then converted to Envarsus Daily (2-5ng/mL) + Everolimus Daily (3-8ng/mL) + prednisone x 6 months
  Interventions: Drug: Tacrolimus; Drug: Prednisone; Drug: Everolimus

INTERVENTIONS:
Drug: Tacrolimus — goal trough level 5-12ng/mL
  Other Names: Envarsus
Drug: Prednisone — goal dose 5mg QD
  Other Names: Corticosteroids; Methylprednisolone
Drug: Mycophenolate mofetil — goal dose 1g BID
  Arms: Tacrolimus + MMF
Drug: Everolimus — goal trough level 3-8ng/mL
  Arms: Envarsus + Everolimus

SUMMARY:
With the availability of well-studied once-daily formulations of tacrolimus, the ability to achieve a true once-daily immunosuppressant regimen along with everolimus and steroids may finally be achievable and have the potential to optimize immunosuppression safety and efficacy in kidney transplantation.

DETAILED DESCRIPTION:
A once-daily immunosuppressant regimen comprising of Envarsus-everolimus-prednisone will have 6-month treatment failure rates that are non-inferior to the twice-daily regimen of Envarsus-mycophenolate mofetil-prednisone and will have improved patient-reported adherence.

ELIGIBILITY:
1. Inclusion criteria

1. Male or female adult (≥18 years old) with a history of solitary kidney transplant within 3 months (±2 months) of transplant with self-reported medication adherence issues, as indicated by a MMAS-8 of at least 1.
2. Patients must be capable of understanding the purposes and risks of the study and have the ability to give written informed consent and be willing to participate and comply with the study.
3. Women of childbearing potential must have a negative pregnancy test within the 48 hours prior to receiving study medication.
4. Women of childbearing potential and sexually active males must be willing to use contraception, as indicated in Section 6 of the protocol. Subjects who are not of reproductive potential (status post bilateral tubal ligation, bilateral oophorectomy, hysterectomy, or vasectomy), not sexually active, whose current partner(s) is not of reproductive potential, or whose sexual activity is exclusively homosexual are eligible without requiring the use of contraception.

2. Exclusion criteria

1. Patients will be excluded if they are pregnant or nursing females or males with a pregnant female partner
2. Recipient of multiple organ transplant
3. Recipient of a non-renal organ
4. Proteinuria > 800 mg/24 hour
5. eGFR < 30 ml/min
6. WBC ≤ 2k/mm3
7. Plt ≤ 50k/mm3
8. Triglycerides > 500 mg/dL
9. HIV positive (HIV ab +)
10. Unable to tolerate oral medications
11. Use of another investigational product within thirty days prior to receiving study medication
12. Acute graft rejection within the past month (Banff 1A or higher) or received an ABO incompatible donor organ.
13. A condition or disorder that, in the opinion of the investigator, may adversely affect the outcome of the study or the safety of the subject

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-12-01 (Actual); Primary Completion 2018-12-27 (Actual); Study Completion 2018-12-27 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

REFERENCES:
- [Derived] Mellon L, Doyle F, Hickey A, Ward KD, de Freitas DG, McCormick PA, O'Connell O, Conlon P. Interventions for increasing immunosuppressant medication adherence in solid organ transplant recipients. Cochrane Database Syst Rev. 2022 Sep 12;9(9):CD012854. doi: 10.1002/14651858.CD012854.pub2. PMID 36094829

RESULTS

PARTICIPANT FLOW:
Groups:
- Control: Envarsus + MMF: Envarsus Daily (5 -12ng/mL) + mycophenolate mofetil 1g BID + prednisone x 6 months
  Tacrolimus: goal trough level 5-12ng/mL
  Prednisone: goal dose 5mg QD
  Mycophenolate mofetil: goal dose 1g BID
- Intervention: Envarsus + Everoliumus: Envarsus Daily (2-5ng/mL) + Everolimus Daily (3-8ng/mL) + prednisone x 6 months
  Tacrolimus: goal trough level 2-5 ng/mL
  Prednisone: goal dose 5mg QD
  Everolimus: goal trough level 3-8ng/mL
Period: Overall Study
Arm/Group | Control: Envarsus + MMF | Intervention: Envarsus + Everoliumus
Started | 20 | 20
Completed | 20 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control: Envarsus + MMF | Intervention: Envarsus + Everoliumus | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.4 (12.9) | 50.3 (14.4) | 51.3 (13.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 6 | 13
  Male | 13 | 14 | 27
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 8 | 10 | 18
  White | 12 | 10 | 22
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Percent of Participants with Medicare Insurance [Count of Participants; unit: Participants] | 14 | 16 | 30
Weight [Mean (Standard Deviation); unit: kg] | 89.7 (15.5) | 88.3 (14.1) | 89.0 (14.6)
Primary Reason for End Stage Renal Disease [Count of Participants; unit: Participants]
  Diabetes | 6 | 7 | 13
  Hypertension | 4 | 5 | 9
  Polycystic Kidney Disease | 2 | 2 | 4
  FSGS | 3 | 1 | 4
  IgA Nephropathy | 2 | 1 | 3
  Lupus | 0 | 1 | 1
  Other | 3 | 3 | 6

OUTCOME MEASURES:

1. Primary Outcome: Self-reported Medication Adherence From Baseline to 6 Months.
Description: Percent of subjects reporting high medication adherence at baseline compared to 6 months post-conversion, using the Morisky Medication Adherence scale (MMAS). The MMAS rates medication adherence on a scale of 0 to 8. 0 is high adherence, 1-2 is medium adherence, and greater than or equal to 3 is low adherence.
Time Frame: 6 months post conversion
Measure: Number; unit: % of participants
Arm/Group | Control: Envarsus + MMF | Intervention: Envarsus + Everoliumus
Number analyzed (Participants) | 20 | 20
% of participants
  Baseline | 80 | 45
  6 months post-conversion | 59 | 47

2. Secondary Outcome: Percent of Participants Experiencing Acute Allograft Rejection
Description: Estimate the composite of treatment failure rate, defined as acute allograft rejection with a Banff grade 1A or higher, graft loss, or death at six months post-conversion, in patients converted to a once-daily immunosuppressant regimen of Envarsus®, everolimus, and prednisone versus patients converted to a twice-daily regimen of Envarsus®, MMF, and prednisone.
Time Frame: Baseline to 6 months post conversion
Measure: Count of Participants; unit: Participants
Arm/Group | Control: Envarsus + MMF | Intervention: Envarsus + Everoliumus
Number analyzed (Participants) | 20 | 20
Participants | 0 | 0

3. Other Pre Specified Outcome: Subject Specific Change on Medication Side Effect Scale
Description: Examine subject specific change on a validated Medication Side Effect Scale at the time of the conversion versus six months post-conversion, compared between the two arms. Side effect burden scale is from 0 to 180. A lower score is less side effect burden, a higher score is more side effect burden.
Time Frame: Baseline to 6 months post conversion
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Control: Envarsus + MMF | Intervention: Envarsus + Everoliumus
Number analyzed (Participants) | 20 | 20
units on a scale
  Baseline | 71 (67) | 37 (38)
  6 month post-conversion | 93 (86) | 38 (34)

4. Other Pre Specified Outcome: Percent of Participants Who Experienced Kidney Transplant Graft Loss
Description: Measure and compare time-to-event analysis between the two arms graft loss (time to event analysis)
Time Frame: Baseline to 6 months post conversion
Measure: Count of Participants; unit: Participants
Arm/Group | Control: Envarsus + MMF | Intervention: Envarsus + Everoliumus
Number analyzed (Participants) | 20 | 20
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: 6 months from Baseline to end of study.
Arm/Group | Control: Envarsus + MMF | Intervention: Envarsus + Everoliumus
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 1/20 | 1/20
Other Adverse Events (participants affected / at risk) | 8/20 | 9/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control: Envarsus + MMF (N=20) | Intervention: Envarsus + Everoliumus (N=20)
JC virus induced Progressive Multifocal Leukoencephalopathy (Infections and infestations) | 1 (1) | 0 (0)
Perinephric fluid collection (Renal and urinary disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control: Envarsus + MMF (N=20) | Intervention: Envarsus + Everoliumus (N=20)
Cytomegalovirus infection (Infections and infestations) | 2 (2) | 1 (1)
Borderline kidney rejection (Renal and urinary disorders) | 1 (1) | 1 (1)
Interstitial Fibrosis and Tubular Atrophy (Renal and urinary disorders) | 2 (2) | 2 (2)
BK infection (Infections and infestations) | 1 (1) | 1 (1)
Lymphocele (Immune system disorders) | 0 (0) | 1 (1)
Diabetic foot ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Neutropenia (Investigations) | 1 (1) | 0 (0)
Graft dysfunction (Renal and urinary disorders) | 0 (0) | 1 (1)
Cardiovascular Event (Cardiac disorders) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-05-11): https://cdn.clinicaltrials.gov/large-docs/98/NCT02954198/Prot_SAP_000.pdf